CLINICAL TRIAL: NCT03215459
Title: CPET-Panc: Exercise Testing in Chemotherapy
Brief Title: Cardiopulmonary Exercise Testing: An Assessment of Patients Fitness for Palliative Chemotherapy for Pancreatic Cancer
Acronym: CPET-Panc
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Collaborators: University of Liverpool Cancer Research Centre (Other)
Responsible Party: Sponsor
Other Study IDs: RDD534
Record Dates: First submitted 2017-06-19; First posted 2017-07-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
Keywords: Cardiopulmonary Exercise Testing
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cardiopulmonary Exercise Test: A cardiopulmonary exercise bike test will be administered prior to palliative chemotherapy treatment.
  Interventions: Device: Cardiopulmonary Exercise Test

INTERVENTIONS:
Device: Cardiopulmonary Exercise Test — Cardiopulmonary Exercise Test

SUMMARY:
Cardiopulmonary exercise testing (CPET) has been shown to be superior to American Society of Anaesthetist classification (ASA) in predicting peri-operative risk. The most common performance status used is the World Health Organisation (WHO) (0-4), with a clinician agreed differentiation of the subsets of 0-2 and 3-4; variability also exists within these subsets.

With this there rises a concern that fit older patients may not be offered appropriate chemotherapy treatment. This observational study will assess whether cardiopulmonary exercise testing (CPET) offers additional benefit over that of WHO Performance status (PS) in the assessment of patients fitness for palliative chemotherapy for pancreatic cancer, by identifying those patients who might survive longer and tolerate chemotherapy better, thus predicting their outcome.

DETAILED DESCRIPTION:
Chemotherapy is widely used to treat a variety of cancers, and is associated with significant complications and even death. The established method for assessing patient fitness is by developing a clinical assessment of patient fitness, and classifying this using a performance status tool. Pancreatic Cancer patients with poorer performance status have been shown to have lower median survival of just 4 months. There is also evidence that patients with poorer performance status have lower response rates to other chemotherapy, higher complication rates, shorter progression free and overall survival. In clinical practice patients with performance status 2 are often offered chemotherapy, even though there is little evidence of its benefit, as the numbers of patients included in clinical trials with PS 2 is low and benefits from chemotherapy appear to be more modest.

Cardiopulmonary exercise testing is a non-invasive test that allows quantification of fitness. It is an objective measure of function capacity/fitness. It has been used in patients due to undergo major surgical intervention, and has the ability to identify those patients who are at higher risk of complications and mortality. CPET has been shown to be superior to the ASA in predicting peri-operative risk. The ASA classification is similar to PS in that it is graded from 1-4, and is a bedside assessment.

Despite the ability of PS to predict outcome it is a fairly blunt tool. The WHO PS is the most commonly used and is graded from 0-4. The categories are broad, for example a WHO PS of 0 could refer to a marathon runner or an elderly patient who is normally relatively inactive. Differentiating between grades is subject to observer error. There is reasonably good agreement between clinicians when differentiating between WHO grade 0-2 and 3-4, however variability exists within these subsets.

More recently it has been noted that it is harder to clinically assess older patients, and there is concern that many fit older patients are not being offered appropriate treatment. This is the subject of a current Department of Health (DoH) equality initiative.

The investigators are interested in identifying whether (CPET) offers additional benefit over that of WHO PS in the assessment of patients fitness for palliative chemotherapy for pancreatic cancer, by identifying those patients who might survive longer and tolerate chemotherapy better, thus predicting their outcome. The CPET variables most commonly used in risk prediction models are the volume of oxygen taken up at the anaerobic threshold relative to body mass (maximal oxygen consumption,VO2 at anaerobic threshold (AT)), the Peak oxygen uptake achieved during the exercise test relative to body mass (VO2 peak) and the oxygen pulse (O2 pulse) which is a derivative value involving oxygen uptake and the heart rate.

The benefit of CPET will be determined by the following:

* Overall survival at 6 months
* Response Rate (Response Evaluation Criteria In Solid Tumors criteria (RECIST) version 1.1)
* 60 day all-cause mortality
* Grade 3 and above adverse events (CTCAE v4) related to chemotherapy
* Chemotherapy dose intensity (% of planned doses given)
* Progression free survival (RECIST criteria version 1.1)
* European Organisation for Research and Treatment of Cancer (EORTC) quality of Life questionnaires (QLQ): to assess quality of life of cancer patients (QLQC30 (version 3)) and participants with pancreatic cancer (QLQ-PAN26)and a health survey 36 questionnaire (RAND 36-item short form health survey 1.0).
* Overall survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven pancreatic cancer
* Due to commence palliative chemotherapy (including as part of a Clinical Trial of an Investigational Medicinal Product (CTIMP)).
* Able to undertake CPET
* Expected life expectancy >3 months
* Age 18+

Exclusion Criteria:

• Haemoglobin <10g/L

Absolute contraindications for cardiopulmonary exercise testing:

* Acute myocardial infarction (3-5 days)
* Unstable angina
* Uncontrolled arrhythmias causing symptoms or hemodynamic comprise
* Syncope
* Active endocarditis
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus or pulmonary infarction
* Thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Room air desaturation at rest ≤85%
* Respiratory failure
* Acute noncardiopulmonary disorder that may aggravated by exercise (i.e. renal failure, thyrotoxicosis)
* Mental impairment leading to inability to cooperate

Relative contraindications for cardiopulmonary exercise testing:

* Left main coronary stenosis or its equivalent
* Moderate stenotic valvular heart disease
* Severe untreated arterial hypertension at rest (>200mm Hg systolic, > 120mm Hg diastolic)
* Tachyarrhythmias or bradyarrhythmias
* High-degree atrioventricular block
* Hypertrophic cardiomyopathy
* Significant pulmonary hypertension
* Advanced or complicated pregnancy
* Orthopaedic impairment that compromises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients from the UK who have Pancreatic cancer and are due to commence palliative chemotherapy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Survival at 6 months (followed up for 12mths) | 6 months
  AUROC (Area under Receiver Operating Characteristic) for WHO (0-4) and WHO + CPET. A logistic regression model will be constructed, one with WHO PS and VO2 at AT (ml/kg/min).
Survival at 6 months (followed up for 12mths) | 6 months
  AUROC for WHO and WHO + CPET: A logistic regression model will be constructed with WHO PS and VO2 max (ml/kg/min).
Survival at 6 months (followed up for 12mths) | 6 months
  AUROC for WHO and WHO + CPET: A logistic regression model will be constructed with WHO PS and O2AT.
Survival at 6 months (followed up for 12mths) | 6 months
  The WHO+CPET classifier with the highest AUROC will then be compared with the AUROC for WHO alone.

SECONDARY OUTCOMES:
Time-to-event endpoints | 6 months
  The Kaplan-Meier method will be used to estimate survival curves.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Palmer, Professor, Principal Investigator — Clatterbridge

IPD SHARING:
Plan to Share IPD: No